CLINICAL TRIAL: NCT05484089
Title: Migration of the CapFlex-PIP Implant System for Proximal Interphalangeal Joint Arthroplasty: a 10 Year Follow up RSA Study
Brief Title: CapFlex PIP Implant RSA
Acronym: Capflex RSA
Status: Recruiting | Type: Observational
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: OC-2021-019
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis Hand
Keywords: RSA; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: CapFlex PIP implant — Patients receive the CapFlex PIP implant based on regular care. During surgery tantalum markers are placed in the bone surrounding the implant.

SUMMARY:
Rationale: Patients with osteoarthrtis (OA) of the proximal interphalangeal (PIP) joint are commonly treated with joint arthroplasty. The CapFlex PIP implant is a modular surface replacing implant, which has good short-term functional results with a relatively low complication rate. To reduce implant failure and to increase long-term survival, it is important to expand knowledge about fixation and loosening patterns. By using model-based roentgen stereogrammaetric analysis (mRSA), the migration pattern of the implant over time can be calculated.

Objective: The primary objective is to assess the fixation and migration patterns of the CapFlex PIP implant system (produced and developed by several companies of KLS Martin Group) in vivo, using mRSA, over 10 years. Secondary objectives are to analyse survival, clinical scores and radiographic aspects of the CapFlex PIP implant system.

Study design: A prospective cohort study with 10 years follow-up, in which 36 patients will be enrolled. Patients will be evaluated preoperatively, at 6 weeks, 6 months, 1 year, 2 years 5 years and 10 years.

Study population: Patients 18 years or older who require a proximal interphalangeal joint arthroplasty as a result of osteoarthritis of a proximal interphalangeal joint.

Main study parameters/endpoints: The main study parameters are the migration of the CapFlex PIP implant system of the distal as well as the proximal component (presented in x-, y- and z-direction). Secondary study parameters are the survival of the CapFlex PIP implant system, clinical scores and radiographic aspects.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients participating in the study will have the same risks when not participating in the study. Patients are asked to spend time to fill in the questionnaires and to have 3 extra visits to the hospital, next to the standard visits. Patients will have more follow up visits and will be followed using RSA analysis, which has as advantage that possible complications might be noticed earlier compared to normal follow up.

ELIGIBILITY:
Inclusion Criteria:

* Indication for PIP joint arthroplasty as described in the manufacturer's guideline, namely as a result of:

  * Painful osteoarthritis
  * Instable communitive intra-articular PIP fractures
* Age > 18 years
* Patient is able to speak and write Dutch
* Patient is willing to participate
* Patient is able and willing to provide written informed consent

Exclusion Criteria:

* Inflammatory arthritis with significant bone loss
* Insufficient bone quality to provide adequate stability
* Known or suspected sensitivity or allergy to one or more of the implant materials
* Revision surgery
* Significant collateral instability
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will get PIP joint arthroplasty.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2035-10 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
The change in Translation in mm | postoperative baseline, 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  Migration will be expressed in the change in translation measured over time compared to the postoperative baseline. Translation is expressed in mm and is given in 3 directions, namely along the x-, y- and z-axes

SECONDARY OUTCOMES:
Rotation in degrees | postoperative baseline, 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  Migration will be expressed in the change in rotation measured over time compared to the postoperative baselin. Rotation is expressed in degrees and is given in 3 directions, namely along the x-, y- and z-axes
Survival | postoperative at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  Survival measured by the percentage of in place implants at each timepoint
Radiographic aspects | postoperative baseline and at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  Radiographic aspects are measured on the x-rays at each time point
Michigan Hand Outcomes Questionnaire (MHOQ) | postoperative baseline and at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  The MHOQ is a validated tool for assessing functional outcome and is divided in six subscales. Each subscale has a formula to calculate a score from 0 (severe disability) to 100 (no disability). The final score is the summation divided by six and goes from 0 (severe disability) to 100 (no disability).
  The MHOQ will be assessed at each time point.
Patient Rated Wrist / Hand Evaluation (PRWHE) | postoperative baseline and at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  The PRWHE measures the patients view on pain, function and cosmetics of the hand/wrist. The maximum score is 150. A high score indicates presence of pain and disability, a low score indicates the absence of pain and disability.
  The PRWHE will be assessed at each time point.
EuroQol-5D (EQ-5D-5L) | postoperative baseline and at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  The EQ-5D-5L is a general health-related quality of life questionnaire. The EQ-5D-5L will be assessed at each time point.
Numeric Rating Scale (NRS) | postoperative baseline and at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years.
  The NRS measures the amount of pain experienced by the patient form 0 (no pain) to 10 (worst pain imaginable).
  The NRS will be assessed at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier Haga Orthopedisch Centrum, Zoetermeer, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided